CLINICAL TRIAL: NCT02141399
Title: A Phase 3 Multicenter Study of the Long-Term Safety and Tolerability of ALKS 5461 for the Adjunctive Treatment of Major Depressive Disorder in Adults Who Have an Inadequate Response to Antidepressant Therapy (the FORWARD-2 Study)
Brief Title: A Long-Term Safety Study of ALKS 5461
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALK5461-208
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — ALKS 5461

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ALKS 5461 (Experimental)
  Interventions: Drug: ALKS 5461

INTERVENTIONS:
Drug: ALKS 5461 — Sublingual tablet, taken daily

SUMMARY:
This is a 52-week open-label study to evaluate the safety and tolerability of ALKS 5461.

ELIGIBILITY:
Inclusion Criteria:

* Agree to use an approved method of contraception for the duration of the study
* Have the potential to safely benefit from the administration of ALKS 5461
* Have a diagnosis of major depressive disorder (MDD)
* Additional criteria may apply

Exclusion Criteria:

* Have a positive test for drugs of abuse
* Currently pregnant or breastfeeding
* Have a current primary Axis-I disorder other than MDD
* Have used opioid agonists (eg, codeine, oxycodone, tramadol, morphine) or opioid antagonists (eg, naloxone, naltrexone) within 14 days
* Have received electroconvulsive therapy treatment within the last 2 years, or received more than 1 course of electroconvulsive treatment during their lifetime
* Have attempted suicide within the past 2 years
* Have a history of intolerance, allergy, or hypersensitivity to buprenorphine or opioid antagonists (eg, naltrexone, naloxone)
* Have had a significant blood loss or blood donation within the past 60 days
* Additional criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1485 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Pathak, MD, Study Director — Alkermes, Inc.
Locations (135):
- United States (108):
  - Alkermes Investigational Site, Birmingham, Alabama
  - Alkermes Investigational Site, Tucson, Arizona
  - Alkermes Investigational Site, Little Rock, Arkansas
  - Alkermes Investigational Site, Bellflower, California
  - Alkermes Investigational Site, Beverly Hills, California
  - Alkermes Investigational Site, Carson, California
  - Alkermes Investigational Site, Garden Grove, California
  - Alkermes Investigational Site, Glendale, California
  - Alkermes Investigational Site, Los Alamitos, California
  - Alkermes Investigational Site, Los Angeles, California
  - Alkermes Investigational Site, National City, California
  - Alkermes Investigational Site, Oakland, California
  - Alkermes Investigational Site, Oceanside, California
  - Alkermes Investigational Site, Orange, California
  - Alkermes Investigational Site, Pico Rivera, California
  - Alkermes Investigational Site, Redlands, California
  - Alkermes Investigational Site, San Gabriel, California
  - Alkermes Investigational Site, Sherman Oaks, California
  - Alkermes Investigational Site, Temecula, California
  - Alkermes Investigational Site, Torrance, California
  - Alkermes Investigational Site, Upland, California
  - Alkermes Investigational Site, Colorado Springs, Colorado
  - Alkermes Investigational Site, Denver, Colorado
  - Alkermes Investigational Site, Hartford, Connecticut
  - Alkermes Investigational Site, Norwich, Connecticut
  - Alkermes Investigational Site, Bradenton, Florida
  - Alkermes Investigational Site, Coral Springs, Florida
  - Alkermes Investigational Site, Fort Myers, Florida
  - Alkermes Investigational Site, Gainesville, Florida
  - Alkermes Investigational Site, Hallandale, Florida
  - Alkermes Investigational Site, Hialeah, Florida
  - Alkermes Investigational Site, Jacksonville, Florida
  - Alkermes Investigational Site, Lauderhill, Florida
  - Alkermes Investigational Site, Maitland, Florida
  - Alkermes Investigational Site, Melbourne, Florida
  - Alkermes Investigational Site, North Miami, Florida
  - Alkermes Investigational Site, Oakland Park, Florida
  - Alkermes Investigational Site, Orlando, Florida
  - Alkermes Investigational Site, Tampa, Florida
  - Alkermes Investigational Site, The Villages, Florida
  - Alkermes Investigational Site, West Palm Beach, Florida
  - Alkermes Investigational Site, Winter Haven, Florida
  - Alkermes Investigational Site, Alpharetta, Georgia
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Decatur, Georgia
  - Alkermes Investigational Site, Smyrna, Georgia
  - Alkermes Investigational Site, Chicago, Illinois
  - Alkermes Investigational Site, Deerfield, Illinois
  - Alkermes Investigational Site, Hoffman Estates, Illinois
  - Alkermes Investigational Site, Joliet, Illinois
  - Alkermes Investigational Site, Oak Brook, Illinois
  - Alkermes Investigational Site, Skokie, Illinois
  - Alkermes Investigational Site, Indianapolis, Indiana
  - Alkermes Investigational Site, Lafayette, Indiana
  - Alkermes Investigational Site, Newburgh, Indiana
  - Alkermes Investigational Site, Valparaiso, Indiana
  - Alkermes Investigational Site, Edgewood, Kentucky
  - Alkermes Investigational Site, Owensboro, Kentucky
  - Alkermes Investigational Site, Baltimore, Maryland
  - Alkermes Investigational Site, Washington D.C., Maryland
  - Alkermes Investigational Site, Belmont, Massachusetts
  - Alkermes Investigational Site, Brockton, Massachusetts
  - Alkermes Investigational Site, Watertown, Massachusetts
  - Alkermes Investigational Site, Worcester, Massachusetts
  - Alkermes Investigational Site, Flowood, Mississippi
  - Alkermes Investigational Site, O'Fallon, Missouri
  - Alkermes Investigational Site, Saint Charles, Missouri
  - Alkermes Investigational Site, St Louis, Missouri
  - Alkermes Investigational Site, Berlin, New Jersey
  - Alkermes Investigational Site, Cherry Hill, New Jersey
  - Alkermes Investigational Site, Princeton, New Jersey
  - Alkermes Investigational Site, Albuquerque, New Mexico
  - Alkermes Investigational Site, Brooklyn, New York
  - Alkermes Investigational Site, Jamaica, New York
  - Alkermes Investigational Site, Mount Kisco, New York
  - Alkermes Investigational Site, New York, New York
  - Alkermes Investigational Site, Staten Island, New York
  - Alkermes Investigational Site, Charlotte, North Carolina
  - Alkermes Investigational Site, High Point, North Carolina
  - Alkermes Investigational Site, Beachwood, Ohio
  - Alkermes Investigational Site, Canton, Ohio
  - Alkermes Investigational Site, Cincinnati, Ohio
  - Alkermes Investigational Site, Dayton, Ohio
  - Alkermes Investigational Site, Mason, Ohio
  - Alkermes Investigational Site, Middleburg Heights, Ohio
  - Alkermes Investigational Site, Oklahoma City, Oklahoma
  - Alkermes Investigational Site, Portland, Oregon
  - Alkermes Investigational Site, Salem, Oregon
  - Alkermes Investigational Site, Allentown, Pennsylvania
  - Alkermes Investigational Site, Media, Pennsylvania
  - Alkermes Investigational Site, Philadelphia, Pennsylvania
  - Alkermes Investigational Site, Lincoln, Rhode Island
  - Alkermes Investigational Site, Charleston, South Carolina
  - Alkermes Investigational Site, Memphis, Tennessee
  - Alkermes Investigational Site, Austin, Texas
  - Alkermes Investigational Site, Dallas, Texas
  - Alkermes Investigational Site, DeSoto, Texas
  - Alkermes Investigational Site, Houston, Texas
  - Alkermes Investigational Site, San Antonio, Texas
  - Alkermes Investigational Site, Sugar Land, Texas
  - Alkermes Investigational Site, Wichita Falls, Texas
  - Alkermes Investigational Site, Clinton, Utah
  - Alkermes Investigational Site, Woodstock, Vermont
  - Alkermes Investigational Site, Bellevue, Washington
  - Alkermes Investigational Site, Seattle, Washington
  - Alkermes Investigational Site, Spokane, Washington
  - Alkermes Investigational Site, Middleton, Wisconsin
  - Alkermes Investigational Site, Waukesha, Wisconsin
- Australia (3):
  - Alkermes Investigational Site, Towong, Queensland
  - Alkermes Investigational Site, Frankston, Victoria
  - Alkermes Investigational Site, Melbourne, Victoria
- Bulgaria (6):
  - Alkermes Investigational Site, Burgas
  - Alkermes Investigational Site, Kazanlak
  - Alkermes Investigational Site, Sofia
  - Alkermes Investigational Site, Varna
  - Alkermes Investigational Site, Veliko Tarnovo
  - Alkermes Investigational Site, Vratsa
- Canada (4):
  - Alkermes Investigational Site, Penticton, British Columbia
  - Alkermes Investigational Site, Halifax, Nova Scotia
  - Alkermes Investigational Site, Gatineau, Quebec
  - Alkermes Investigational Site, Québec
- Germany (9):
  - Alkermes Investigational Site, Oranienburg, Brandenburg
  - Alkermes Investigational Site, Achim
  - Alkermes Investigational Site, Berlin
  - Alkermes Investigational Site, Ellwangen
  - Alkermes Investigational Site, Freiburg im Breisgau
  - Alkermes Investigational Site, Hanover
  - Alkermes Investigational Site, Mainz
  - Alkermes Investigational Site, Schwerin
  - Alkermes Investigational Site, Stralsund
- Alkermes Investigational Site, Budapest, Hungary
- Poland (3):
  - Alkermes Investigational Site, Bialystok
  - Alkermes Investigational Site, Gdansk
  - Alkermes Investigational Site, Gorlice
- Alkermes Investigational Site, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were entered into the study in one of 3 ways, based upon previous experience with a prior ALKS 5461 study: Subjects continuing from a prior ALKS 5461 study; Subjects who participated in the prospective lead-in for a prior ALKS 5461 study, but did not meet the entrance criteria; Subjects who did not participate in a prior ALKS 5461 study.
Pre-assignment Details: All subjects received ALKS 5461 during the course of the study as an adjunctive treatment for major depressive disorder. In addition all subjects were treated with background antidepressant therapy prescribed by the investigator.
Groups:
- ALKS 5461: ALKS 5461 adjunctive treatment
Period: Overall Study
Arm/Group | ALKS 5461
Started | 1485
Completed | 741
Not Completed | 744
Not completed — Adverse Event | 158
Not completed — Lack of Efficacy | 62
Not completed — Lost to Follow-up | 151
Not completed — Non-compliance with study drug | 18
Not completed — Other | 45
Not completed — Physician Decision | 17
Not completed — Pregnancy | 3
Not completed — Protocol Violation | 38
Not completed — Withdrawal by Subject | 238
Not completed — Failure to meet eligibility criteria | 14

BASELINE CHARACTERISTICS:
Population: The safety population includes all subjects who received at least 1 dose of study drug.
Arm/Group | ALKS 5461
Number analyzed (Participants) | 1485
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 964
  Male | 521
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 197
  Not Hispanic or Latino | 1288
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7
  Asian | 28
  Native Hawaiian or Other Pacific Islander | 8
  Black or African American | 362
  White | 1080
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 54
  Hungary | 5
  United States | 1204
  Poland | 33
  Australia | 35
  Bulgaria | 88
  Germany | 66

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events (AEs)
Time Frame: Up to 56 weeks
Population: The safety population included all subjects who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ALKS 5461
Number analyzed (Participants) | 1485
Participants | 1124

ADVERSE EVENTS:
Time Frame: Up to 56 weeks
Arm/Group | ALKS 5461
All-Cause Mortality (participants affected / at risk) | 2/1485
Serious Adverse Events (participants affected / at risk) | 47/1485
Other Adverse Events (participants affected / at risk) | 1124/1485
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALKS 5461 (N=1485)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Depression (Psychiatric disorders) | 3 (3)
Suicidal ideation (Psychiatric disorders) | 3 (3)
Colitis (Gastrointestinal disorders) | 2 (2)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Myocardial infarction (Cardiac disorders) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Meningitis viral (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral Haemorrhage (Nervous system disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Major depression (Psychiatric disorders) | 2 (2)
Conversion disorder (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALKS 5461 (N=1485)
Nausea (Gastrointestinal disorders) | 322 (409)
Constipation (Gastrointestinal disorders) | 151 (173)
Vomiting (Gastrointestinal disorders) | 116 (134)
Dry mouth (Gastrointestinal disorders) | 87 (95)
Headache (Nervous system disorders) | 156 (198)
Dizziness (Nervous system disorders) | 150 (179)
Somnolence (Nervous system disorders) | 124 (142)
Upper respiratory tract infection (Infections and infestations) | 83 (98)
Nasopharyngitis (Infections and infestations) | 80 (88)
Insomnia (Psychiatric disorders) | 81 (90)
Fatigue (General disorders) | 85 (91)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should an Investigator desire to disclose study results, Sponsor will review the results disclosure prior to public release and can embargo the disclosure for a period of at least 60 days. Revisions to the disclosure will be negotiated in good faith. For a multicenter study the Investigators agree to publish/publicly present the results together with the other sites for the 12 month period after study results are available unless Sponsor grants written permission in advance.

DOCUMENTS (2):
  • Study Protocol (2016-03-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT02141399/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT02141399/SAP_001.pdf